CLINICAL TRIAL: NCT05567536
Title: HOST-EXAM-Ex : Harmonizing Optimal Strategy for Treatment of Coronary Artery Stenosis - EXtended Antiplatelet Monotherapy - EXtended Follow up
Brief Title: Long Term Follow-up of Comparison of Clopidogrel vs. Aspirin Monotherapy After Drug-eluting Stent Implantation
Acronym: HOST-EXAM-EX
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Department of Internal Medicine, Seoul National University Hospital
Other Study IDs: 1208-028-421
Record Dates: First submitted 2022-09-26; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; Atheroscleroses, Coronary
Keywords: percutenous coronary intervention; drug-eluting stent; chronic maintenance period
MeSH Terms: conditions — Coronary Artery Disease | interventions — Platelet Aggregation Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clopidogrel group: This group are those who received clopidogrel 75mg qd as a single antiplatelet agent therapy after PCI.
  Interventions: Drug: Antiplatelet Agents
- Aspirin group: This group are those who received aspirin 100mg qd as a single antiplatelet agent therapy after PCI.
  Interventions: Drug: Antiplatelet Agents

INTERVENTIONS:
Drug: Antiplatelet Agents — Patients who received a single antiplatelet agent will be analyzed according to the prescribed antiplatelet agent

SUMMARY:
This is an retrospective extended study of a randomized clinical trial (The HOST-EXAM trial ClinicalTrials.gov Identifier: NCT02044250).

Investigators will perform a retrospective analysis of all participants enrolled in this trial will be performed, until the longest follow-up duration.

DETAILED DESCRIPTION:
The HOST-EXAM trial (ClinicalTrials.gov Identifier: NCT02044250) was an randomized clinical trial that was performed to compare head-to-head, the efficacy and safety between aspirin and clopidogrel monotherapy in patients who received PCI for coronary artery disease and required chronic maintenance antiplatelet therapy. From March 2014 through May 2018, a total of 5438 patients were enrolled, and follow-up was performed upto 24 months after randomization. After this study, randomization was unlocked and patients were followed-up based on the standard protocol.

Afterwards, the current study was planned to perform a extended follow-up of the HOST-EXAM population. The specific drug by the randomization group in the HOST-EXAM trial was not mandatory after the initial 24 months, therefore participants received medication according to the current guidelines, and according to the physicians preferences.

This is a observational, retrospective analysis of all clinical events after the randomization period. The prescribed medications and any clinical events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were enrolled in the HOST-EXAM randomized clinical trial

Exclusion Criteria:

* None, otherwise the patient refuses to participate in this study, or refuses to provide personal medical information

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were enrolled in the HOST-EXAM randomized clinical trial will be analyzed for an extended follow-up duration.
  Patients enrolled in the HOST-EXAM trial were patients that received stenting with a drug-eluting stent and had successfully completed 6-18 months of DAPT without events.
Sampling Method: Non-Probability Sample
Enrollment: 5530 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient oriented composite outcome | From date of randomization until March, 2022.
  A composite of all-cause death, nonfatal myocardial infarction, stroke, readmission due to acute coronary syndrome, and major bleeding complication

SECONDARY OUTCOMES:
Thrombotic outcome | From date of randomization until March, 2022.
  cardiac death, non-fatal MI, ischemic stroke, readmission due to ACS, and definite or probable stent thrombosis
Bleeding outcome | From date of randomization until March, 2022.
  Bleeding Academic Research Consortium (BARC) type ≥2 bleeding

OTHER OUTCOMES:
All-cause death | From date of randomization until March, 2022.
  Death from any cause
Cardiac death | From date of randomization until March, 2022.
  Death from a cardiac cause

IPD SHARING:
Plan to Share IPD: No
The HOST-EXAM-Ex study is planning to continue follow-up until 2028. No individual participant data will be available before this. Any relevant inquiries should be sent to the central contact person or backup person.

REFERENCES:
- [Result] Koo BK, Kang J, Park KW, Rhee TM, Yang HM, Won KB, Rha SW, Bae JW, Lee NH, Hur SH, Yoon J, Park TH, Kim BS, Lim SW, Cho YH, Jeon DW, Kim SH, Han JK, Shin ES, Kim HS; HOST-EXAM investigators. Aspirin versus clopidogrel for chronic maintenance monotherapy after percutaneous coronary intervention (HOST-EXAM): an investigator-initiated, prospective, randomised, open-label, multicentre trial. Lancet. 2021 Jun 26;397(10293):2487-2496. doi: 10.1016/S0140-6736(21)01063-1. Epub 2021 May 16. PMID 34010616
- [Result] Antithrombotic Trialists' (ATT) Collaboration; Baigent C, Blackwell L, Collins R, Emberson J, Godwin J, Peto R, Buring J, Hennekens C, Kearney P, Meade T, Patrono C, Roncaglioni MC, Zanchetti A. Aspirin in the primary and secondary prevention of vascular disease: collaborative meta-analysis of individual participant data from randomised trials. Lancet. 2009 May 30;373(9678):1849-60. doi: 10.1016/S0140-6736(09)60503-1. PMID 19482214